CLINICAL TRIAL: NCT02567214
Title: Indacaterol 110µg/ Glycopyrronium 50µg (Ultibro®) Versus Tiotropium (Spiriva®) Alone to Reduce Exertional Dyspnea in Patients With Moderate to Severe COPD
Brief Title: Ultibro® Versus Spiriva® Alone to Reduce Exertional Dyspnea in Patients With Moderate to Severe COPD
Acronym: RED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Francois Maltlais, MD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-10-2016-2572
Record Dates: First submitted 2015-09-25; First posted 2015-10-02 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: COPD
Keywords: dyspnea; exercise; shuttle test; long-acting β2-agonists; longacting muscarinic antagonist; indacaterol; glycopyrronium; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity | interventions — indacaterol; Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultibro® versus sham Spiriva® (Experimental): Indacaterol 110 µg/Glycopyrronium 50 µg Inhaled
  1 time per day 21 days
  Interventions: Drug: Ultibro®
- Sham Ultibro® versus Spiriva® (Experimental): Tiotropium 18 µg Inhaled
  1 time per day 21 days
  Interventions: Drug: Spiriva®

INTERVENTIONS:
Drug: Ultibro® — The intervention in this arm is the Ultibro®. To keep the patients blinded on which treatement they are taking they will use the two devices but in this arm the Ultibro will be delivered and the Spiriva will be a placebo. We will measure the exertional dyspnea after 21 days of treatment.
  Other Names: Indacaterol 110 µg/Glycopyrronium 50 µg
  Arms: Ultibro® versus sham Spiriva®
Drug: Spiriva® — The intervention in this arm is the Spiriva®. To keep the patients blinded on which treatement they are taking they will use the two devices but in this arm the Ultibro will be a placebo and the Spiriva will be delivered. We will measure the exertional dyspnea after 21 days of treatment.
  Other Names: Tiotropium 18 µg
  Arms: Sham Ultibro® versus Spiriva®

SUMMARY:
The investigators will compare the reduction in Borg dyspnea score during the 3-min constant rate shuttle walking test after 3 weeks of indacaterol 110 µg/Glycopyrronium 50 µg (Ultibro®) versus Tiotropium 18 µg (Spiriva®) alone in patients with moderate to severe COPD.

DETAILED DESCRIPTION:
The foundation of COPD therapy is to combine inhaled therapy to optimize benefits as it was done several years ago by associating short-acting β2-agonists and muscarinic antagonist. The recent availability of once-daily LABA/LAMA fixed combination products makes this therapeutic strategy even more appealing and appears as a promising treatment option in COPD. One relevant question regarding these new LABA/LAMA combinations is whether they provide superior benefits compared to a single agent. Once-daily LABA/LAMA fixed combinations consistently improves lung function compared to monotherapy. The key question is whether they provide superior efficacy to monotherapy on patient's oriented clinical outcomes, beyond lung function improvement. In regards, once-daily LABA/LAMA fixed combinations can reduce exacerbation rate and perception of dyspnea, further to what can be obtained with the monocomponents. Once-daily LABA/LAMA fixed combinations also improve exercise tolerance compared to placebo but whether they provide additional benefit over monotherapy is uncertain.

Dyspnea is the most troublesome symptom in COPD and it is felt that the main mechanism through which bronchodilators improve exercise tolerance is by reducing dyspnea. As such, dyspnea measurement appears a valid surrogate of exercise tolerance. One advantage of dyspnea measurement over the measurement of exercise endurance is that it does not require a maximal effort. In this regard, it may be a less noisy outcome than exercise duration. Dyspnea can be quantified during the 6-min walking test but pre and post-intervention comparisons are made difficult since the walking speed and thus the exercise stimulus is not controlled during the test. Another strategy to evaluate the effects of interventions on exertional dyspnea is to compare dyspnea at isotime while controlling the walking or cycling speed during the endurance shuttle walking test or the constant rate cycling test. One limitation of this approach is that pre and post intervention dyspnea measurement is not always obtained at the same time point since the duration of the test is variable. To overcome this problem, linear interpolation can be used to estimate of dyspnea. However, this approach is not as robust as when a "real" dyspnea score is directly obtained from the patients.

To circumvent these difficulties, the investigators have recently developed a strong and simple exercise methodology whose primary objective is to assess exertional dyspnea in patients with COPD: the 3-min constant rate shuttle walking test. During this test, which is a modification of the endurance shuttle walking test, patients are asked to walk around two cones set-up in a flat corridor and separated by 10m. An audio signal is used to impose the walking speed and the test ends at a fixed duration of 3 minutes or until symptoms become intolerable. At pre-specified time point during the test, and at the end of the test (3 min), patients are asked to score their perception of dyspnea on a Borg scale. The feasibility and reproducibility of this test in providing a standardized physical stimulus and a measurable level of dyspnea in patients with moderate to severe COPD has been reported. In one study, the investigators also confirmed the responsiveness of this test to bronchodilation, reporting statistically and clinically significant reduction in Borg dyspnea score with ipratropium bromide compared to placebo.

Methodology:

The study will require 7 visits; the run-in and familiarization phase (visits #1-3), the treatment A phase (visits #4-5), and the treatment B phase (visits #6-7).

The first visit will be used to review the inclusion criteria and to obtain consent. A spirometry will be obtained. Patient on tiotropium or glycopyrronium will be switched to open label ipratropium (see allowed medication). Visit #2 will include pulmonary function testing including spirometry, lung volumes and diffusion capacity measurements. A maximal incremental shuttle walking test, the COPD assessment test (CAT) and the MRC scale will be also be completed. Patients will then be familiarized with the 3-min constant rate shuttle walking test. During Visit #3, patients will perform two 3-min constant rate shuttle walking test which will serve to determine dyspnea at baseline. The investigators will aim for a dyspnea Borg Score > 3, the rationale being that it is important to obtain a significant dyspnea signal considering that the objective of the study is to evaluate the efficacy of bronchodilation to improve dyspnea. Patients in whom it will not be possible to achieve this level of dyspnea at the end of the 3- min constant rate shuttle walking test will be excluded for further study participation.

Patients will then enter the cross-over study design during which they will receive one of the two study treatments: indacaterol 110 µg/Glycopyrronium 50 µg (Ultibro®) once a day or Tiotropium 18 µg (Spiriva®) once a day. The treatment period will be three weeks. There will be a 2-week washout period between the two treatment phases. Total study duration will thus be 11 weeks.

Visit #4 and visit #6 will be the baseline visits for each treatment period (except for dyspnea after the 3-min constant rate shuttle walking test which will be determined at Visit #3). Participants will perform spirometry, lung volume measurements before and 1h 20 min after receiving the study medication. Two 3-min constant rate shuttle walking tests will be performed 2h 25 min after dosing, starting with the one performed and completed at the highest speed at V3. This time schedule was chosen based on previous studies in this field. Dyspnea will be assessed with the baseline dyspnea index (BDI) and health status will be evaluated by the COPD Assessment Test (CAT).

The same procedures will be repeated at the end of each 3-week study treatment (Visits #5 and #7) the only difference being that chronic dyspnea will be assessed with the transitional dyspnea index (TDI).

Allowed medication There will be a 3-week run-in period during which patients on will receive open label ipratropium (Atrovent® MDI 20µg/ puff, 4 puffs QID) and prn salbutamol (Ventolin® MDI 100µg/puff, 2 puffs every 3-4 hours PRN). Ipratropium will be allowed only during the run-in and washout periods. Ipratropium will be stopped twelve hours before study visits (Visit # 3, 4, and 6).

Salbutamol on prn basis will allow throughout the study except that it will be stopped 6 hours prior to Visit #3, 4, 5, 6 and 7. Long-acting 2-agonist will be prohibited after Visit #1 and throughout study duration. Inhaled corticosteroids will be allowed at the same dosage as before the study. PDE4 inhibitors and leukotriene antagonists will also be allowed.

Blinding Patient and study staff will be blinded to the treatment administration during the 2 study periods. Treatments will consisted, for one treatment period of active Ultibro® once a day and placebo Spiriva® handihaler, and for the other period of placebo Ultibro® once a day and active Spiriva® handihaler. Active medication and placebo will be of identical appearance and the order of study medication will be randomized. Pre-package envelopes containing equal quantities of inhaler combination will be numbered and kept in a secure place (pharmacy of the hospital or the research site). At the end of the study data collection the blind code will be opened after having completed the primary data analysis.

Randomization stratified by site will occur at Visit #4 and will be centralized using a computerized system and pre-packaged study medication.

Evaluation criteria:

Primary endpoint will be the difference in Borg dyspnea score after the 3-min constant rate shuttle walking test after 3 weeks of treatment between indacaterol 110µg/Glycopyrronium 50µg (Ultibro®) versus Tiotropium 18µg (Spiriva®) alone. Secondary endpoints will be the difference in Borg dyspnea score after the 3-min constant rate shuttle walking test after 3 weeks of treatment between indacaterol 110µg/Glycopyrronium 50µg (Ultibro®) versus baseline value (Visit #3) and between Tiotropium 18µg (Spiriva®) alone versus baseline value (Visit #3). The dyspnea response after the first dose of therapy will also be assessed. The between-treatment differences in the improvement of pulmonary function (FEV1 and inspiratory capacity), TDI and CAT scores from baseline (V4) to end of treatment period (V5 and V7) will also be evaluated.

Assessment and procedures

Pulmonary function testing. Spirometry, lung volumes and diffusion capacity will be measured according to routine techniques.

Maximal incremental shuttle walk. As originally described by Singh and colleagues, the incremental shuttle walk will be performed in an enclosed corridor on a flat 10-m-long course. The course will be identified by two cones, each positioned 0.5 m from either end to allow patients to walk in circle and thereby avoid the need for abrupt changes in direction. Patients will walk at a predetermined rhythm, as dictated by an audio signal played from a CD. Walking speed will initially be set at 0.50 m/sec and will be increased by 0.17 m/sec every minute until the patient reaches maximal capacity. Since the effects of encouragement on walking performance have been demonstrated, no encouragement will be given to patients throughout the test. The final measure will be distance walked, expressed in meters.

3-min constant rate shuttle walking test. This test consists in one bout of three minutes of walking at the initial walking speed of 4.0 km/h. Thirty minutes after this first bout of walking, a second test will be performed at a walking speed of either 6.0 or 2.5 km/h. The second walking speed will be determined by the ability to carry through the test at 4.0 km/h. If a patient cannot complete the first test, then the second speed will be stepped down to 2.5 km/h. If a patient is able to carry though the first test, then the second walking speed will be raised to 6.0 km/h. Patients will be asked to perform two tests at two different speeds in order to determine, amongst the 3 different walking speeds, the highest speed that can be sustained for the entire 3 minutes. In doing so, our objective is to induce a level of dyspnea that is sufficiently high to be amenable to therapy. These walking speeds are selected based on our previous work19 showing that these were sufficiently demanding to induce measurable levels of dyspnea and that most moderate to severe patients with COPD are able to complete the test for the desired duration. Patients will be directed to follow the audio signal for the entire 3 minutes of the test or until they became symptom limited. They will be instructed to walk around the two cones set-up in the hospital hallway pacing their walk in a way not to wait at the cones for the following audio signal.

Cardiac and ventilatory measures. During each exercise test, cardiac and ventilatory parameters will be measured using a commercially available exercise circuit. Dyspnea will be assessed using a 10-point modified Borg scale that will be positioned at one extremity of the course.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Smoking history > 10 packs/year
3. FEV1 30 - 79% of predicted and FEV1/FVC < 70% (GOLD 2-3)
4. FRC > 120 % predicted
5. Borg dyspnea score > 3 during the 3-min constant rate shuttle walking test at V3

Exclusion Criteria:

1. Respiratory exacerbation within the 2 months preceding the study
2. Current diagnostic of asthma
3. Significant O2 desaturation (SpO2 < 85%) at rest or during exercise
4. Presence of another pathology that could influence exercise tolerance
5. Use of home oxygen

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Reduction of dyspnea score during the 3-min constant rate shuttle walk test | 21 days
  To compare the reduction in dyspnea in each arm of the study using the BORG scale and the questionnaire BDI-TDI.

SECONDARY OUTCOMES:
Improvement of the pulmonary function after taking Ultibro® and Spiriva® | 21 days
  To compare the effect of the two treatments on the pulmonary function measured by plethysmography.
Impact of Ultibro® and Spiriva® on exertional dyspnea after the first dose of therapy | 1 day
  We will assess the dyspnea, using the BORG scale during the 3-min constant rate shuttle walk test (CRSWT). The CRSWT will be done after the patient receive the first dose in each arm of the study.
Impact of Ultibro® and Spiriva® on quality of life measured with the CAT questionnaire. | 21 days
  To compare the effect of the two treatments on the quality of life measured by the CAT questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University
Locations (3):
- Canada (3):
  - Queens University, Kingston, Ontario
  - McGill University, Montreal, Quebec
  - Laval University - IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02567214/Prot_000.pdf